CLINICAL TRIAL: NCT06154616
Title: Analysis of the Efficacy of Different Types of Milk Enriched With Tryptophan and Supplemented With Ashwagandha Extract in Improving Sleep Quality in Subjects With Sleep Problems
Brief Title: Efficacy of Different Types of Milk in Improving Sleep Quality in Subjects With Sleep Problems (Milca)
Acronym: Milca
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UCAMCFE-00033
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-09

CONDITIONS: Poor Quality Sleep
Keywords: Ashwagandha extract; tryptophan
MeSH Terms: interventions — Control Groups; tryptophyltryptophan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): Subjects will consume 250 ml of milk half an hour before bedtime.
  Interventions: Dietary Supplement: Control Product
- Ashw 250 (Experimental): Subjects will consume 250 ml of milk half an hour before bedtime.
  Interventions: Dietary Supplement: Experimental Product: 250
- Ashw 250 + TRP (Experimental): Subjects will consume 250 ml of milk half an hour before bedtime.
  Interventions: Dietary Supplement: Experimental Product: 250 + TRP
- Ashw 600 (Experimental): Subjects will consume 250 ml of milk half an hour before bedtime.
  Interventions: Dietary Supplement: Experimental Product: 600

INTERVENTIONS:
Dietary Supplement: Control Product — Lactose-free skimmed milk
  Arms: Control
Dietary Supplement: Experimental Product: 250 — Lactose-free skimmed milk enriched with 250 mg aswaghanda
  Arms: Ashw 250
Dietary Supplement: Experimental Product: 250 + TRP — Lactose-free skimmed milk enriched with 250 mg aswaghanda and tryptophan
  Arms: Ashw 250 + TRP
Dietary Supplement: Experimental Product: 600 — Lactose-free skimmed milk enriched with 600 mg aswaghanda
  Arms: Ashw 600

SUMMARY:
Randomized, controlled, double-blind intervention study, with four parallel branches depending on the product consumed, to analyze the efficacy of different types of milks on the improvement of sleep quality.

DETAILED DESCRIPTION:
The duration of the study will be 90 days (12 weeks). Each day they will have to consume the product under investigation. The subjects who meet the selection criteria will be randomly distributed in each of the study groups (A, B, C or D, depending on the group in which they have been randomized). Each day the subjects will have to fill in a diary on sleep quality and concomitant medication.

They will make a total of two visits to the research laboratory and the tests preestablished in the protocol will be performed. Subsequently, a statistical analysis will be performed with the variables measured in the study to obtain the results.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (> 18 years).
* Low sleep quality by Pittsburgh Sleep Quality Questionnaire (PSQI).
* Volunteers able to understand the clinical study and willing to comply with the study procedures and requirements.

Exclusion Criteria:

* Subjects with serious or terminal illnesses.
* Subjects with known allergy or hypersensitivity to any of the components of the investigational product.
* Participation in another study involving blood draws or dietary intervention.
* Subjects with body mass index above 32 kg/m2.
* Pregnant or lactating women.
* Use of medications that alter cognitive functions or sleep, such as barbiturates, anticonvulsants, benzodiazepines, antidepressants, neuroleptics, alcohol and illicit drugs.
* Organic dementias such as Alzheimer's, Huntington's disease, Parkinson's and senile dementia.
* Inability to understand informed consent (IC).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Variation in sleep quality from baseline at 12 weeks. | The evolution of sleep quality after consumption during 12 weeks will be measured.
  Visual analog scale from 0 to 10. The higher the value, the more quality.

SECONDARY OUTCOMES:
Change in Sleep Quality from baseline at 12 weeks | Sleep quality will be measured with a daily scale, from baseline to 12 weeks.
  Visual analog scale from 0 to 10. The higher the value, the more quality.
Sleep quality | It will be measured twice, once at baseline or at the end of the study after 12 weeks of use
  Measured by Pittsburgh test
Insomnia severity | It will be measured twice, once at baseline or at the end of the study after 12 weeks of use
  Measured by Insomnia severity index - ISI test
Sleepiness | It will be measured twice, once at baseline or at the end of the study after 12 weeks of use
  Measured by Epworth test
Matutinity - Verpertinity | It will be measured twice, once at baseline or at the end of the study after 12 weeks of use
  Measured by Matutinity - Verpertinity questionnaire
Anxiety questionnaire | Day 1, at 12 weeks later
  Test STAI, to measure the level of anxiety of the subjects
Body composition | The test will be measured at baseline and after 12 weeks of consumption.
  It is a control variable. Measured by bioimpedance
Adverse events | At 12 weeks after consumption
  It will be evaluated at each of the visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain